CLINICAL TRIAL: NCT04254393
Title: Early Adolescent Skills for Emotions (EASE) - A Skills Based Program to Address Psychosocial Distress Among Young Adolescents Studying in Public Schools of Pakistan. Pilot Cluster Randomized Controlled Trial (cRCT)
Brief Title: Early Adolescent Skills for Emotions (EASE)-Pilot Cluster Randomized Controlled Trial (cRCT) in Public Schools of Rural Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: University of Liverpool (Other); Institute of Psychiatry, WHO Collaborating Center for Mental Health, Rawalpindi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EASE Pilot cRCT
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Psychological Distress; Emotional Problem; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — methyl hydroxyethyl cellulose; Therapeutics

STUDY DESIGN:
Intervention Model Description: Two arm, single blind, pilot cluster randomized controlled trial (cRCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators and outcome assessors will be blind to the allocations status of participants. To ensure blinding, participants will be instructed to not disclose their allocation during assessment.
  Fidelity of masking will be ensured by having assessors guess the allocation status of participants at the end of assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Adolescent Skills for Emotions (EASE) Program (Experimental): Early Adolescent Skills for Emotions (EASE) is a new, brief, targeted, group psychological intervention program (Dawson et al., 2019) based on cognitive behavioural therapy (CBT) techniques that are empirically supported and formally recommended by the WHO (WHO, 2016).
  Interventions: Behavioral: Early Adolescent Skills for Emotions (EASE) Program
- Treatment as Usual (TAU) (Placebo Comparator): Participants in control arm will be able to avail the routine services available in school settings.
  Interventions: Other: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Early Adolescent Skills for Emotions (EASE) Program — EASE has been developed to manage and reduce symptoms of depression, anxiety and distress in adolescents. EASE is designed to be delivered by non-specialists in low resource settings such as a trained school-health counsellor. The intervention comprises of 7 young adolescent group sessions, each lasting 90 minutes and involves the empirically supported components of psycho education, problem solving, stress management (slow breathing), behavioural activation, and relapse prevention and 3 caregiver group sessions, each lasting 120 minutes and involve psycho education, active listening, quality time, praise, caregiver self-care and relapse prevention.
  Arms: Early Adolescent Skills for Emotions (EASE) Program
Other: Treatment As Usual (TAU) — Evidence based health practices are not available in schools to manage the mental health problems of children. No structured programs are being implemented in school settings for at-risk children. During the study, participants in TAU showing severe psychiatric symptoms that require immediate specialist treatment and follow-up, will be referred to the Institute of psychiatry (IoP)-the tertiary mental health care facility of the region.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Background: Emotional problems such as symptoms of depression, anxiety and psychosocial distress are the leading contributors to health burden among adolescents worldwide. There is an urgent need for evidence-based psychological interventions for young people, especially those living in adversity. WHO has developed Early Adolescent Skills for Emotions (EASE), a brief group psychological intervention delivered by non-specialist providers for young adolescents impaired by distress and exposed to adversity. We aim to evaluate the feasibility of delivering EASE for young adolescents living in public schools of rural Rawalpindi, Pakistan.

Objectives: To evaluate the feasibility of delivering Early Adolescent Skills for Emotions (EASE) program to young adolescents and their caregivers in Rawalpindi, Pakistan to inform the design, including sample size estimation, for a full-scale adequately powered definitive cluster randomised controlled trial.

Methods: A two arm, single blind, pilot cluster randomized controlled trial will be conducted with adolescents of both gender (aged 13-15 years) with high psychological distress, studying in grade 8 and 9th of middle and high public school in rural Rawalpindi.

Schools will be the units of randomization. 8 public schools, stratified by gender, will be randomized into EASE plus Treatment as Usual (TAU) (n=4) and TAU alone (n=6). 60 young adolescents at-risk of psychosocial distress as assessed by Self-Reported-Pediatric Symptom Checklist (PSC), cut-off ≥28 will be included in the study. No power calculations have been calculated for the present pilot trial; however, the sample will be adequate to inform the parameters of planned definitive cRCT. In the intervention arm, adolescents will receive 7-weekly group sessions and their caregivers will receive 3-weekly group sessions in public schools. Data on the number of outcomes will be collected at baseline, immediately and 3-months' post-intervention follow-up. The findings will inform the sample size required for a definitive trial. A detailed mixed-methods process evaluation will be conducted to identify areas of improvements prior to proceeding to a definitive cRCT.

Discussion: The results of pilot trial will be used to inform the design of definitive cluster randomized controlled trial in government led scaled-up implementation of healthy school initiative in Rawalpindi district of Pakistan.

ELIGIBILITY:
The study participants will be 60 adolescents (aged 13-15), at-risk of psycho-social distress as assessed by self-reported Pediatric Symptoms Check list (score ≥ 28); studying in public schools of rural Rawalpindi, Pakistan and their primary caregivers. To estimate the magnitude of treatment effect and its variation for a sample size calculation in the definitive trial, a pilot study sample size of 24 - 50 has been recommended (Browne, 1995; Julious 2005). With a sample size of 60 (30 per arm), we aim to generate some reliable estimate of treatment effect as well as recruitment and attrition rates.

Adolescents in need of acute protection (at high risk of abuse or harm to self or others) and who require immediate or ongoing medical or psychiatric care reported by parents will be excluded from the study.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Symptoms Checklist (PSC) | At 3-months' post-intervention.
  Self-rated Pediatric Symptom Checklist (PSC) will be used to assess psychosocial distress of adolescents. Pediatric symptom checklist has 35 items and assesses psychosocial problems on 3 subscales; externalizing, internalizing and attention problems with cut-offs of 7, 5, 7 respectively. Items are rated on a three-point Likert scale (0= Never, 1= Sometimes, 2=Often). Total score is calculated by summing the responses of all items. Higher score indicates greater psychosocial distress. The recommended cutoff for identifying children and adolescents with psychosocial distress using Pediatric Symptom Checklist in a new setting is ≥ 28.

SECONDARY OUTCOMES:
Somatic-symptom questionnaire | At baseline, immediate and 3-months' post-intervention.
  The somatic symptoms questionnaire will be used to measure stress management among adolescents. It consists of 10 items, rated on a 3-point scale (0=not true, 1=somewhat true, 2= very true or often true) based on the occurrence of the symptoms. Total score is calculated by summing the responses of all items. Higher score indicates frequent occurrence of somatic symptoms.
Social Problem-Solving Inventory - Revised Short Form | At baseline, immediate and 3-months' post-intervention.
  It is a self-reporting questionnaire with 25 items. It consists of five sub-scales with five items each. Two of these sub-scales, 'positive problem orientation' and 'negative problem orientation', assess functional and dysfunctional cognitive and emotional orientations towards solving problems. The three remaining sub-scales, 'rational problem solving', 'impulsivity-carelessness style', and 'avoidance style', assess problem-solving skills and behavioral style. The total score of this scale varies between 0 and 20 points. Highest scores correspond to better social problem-solving abilities.
Perceived Emotional/Personal Support Scale | At baseline, immediate and 3- months' post-intervention.
  It assesses perceived emotional support. Respondents are instructed to list the gender and first initial of three important people in each of three relationship categories: family members, non-family adults, and friends. Using a four-point scale (hardly at all to very much), respondents answer the following questions about each person listed: "How much do you talk to them about personal concerns?" "How close do you feel to them?" and "How satisfied are you with the help and support they give you?" How much do they talk to you about their concerns? Three support variables are created by averaging all ratings for all persons listed within each relationship category: perceived support from family, non-family adults, and peers. Scores range from 1 to 4.
Patient Health Questionnaire (PHQ-9)- adapted for adolescents | At baseline, immediate and 3-months' post-intervention.
  PHQ-9, adapted for adolescents will be used to assess depression symptoms and severity among adolescents. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. It is used to monitor the severity of depression and response to treatment. Items are rated on a 4-point Likert scale with 0= Not at all, 1= Several Day, 2= More than half the days, 3= nearly every day. Total score is calculated by summing the responses of all items. Higher score indicates higher incidence of depression symptoms. PHQ-9 total score for the nine items ranges from 0 to 27. PHQ-9 scan also be used to screen presence of depressive symptoms in adolescents; where score 0-4 indicates 'absence of depressive symptoms', score 5-9 indicates 'mild depression', score 10-14 indicates 'moderate depression', 15-19 indicates 'moderately severe depression', score 20-27 indicates presence of 'severe depression'.
Pediatric Quality of Life (PedsQL) | At baseline, immediate and 3-months' post-intervention.
  Pediatric Quality of Life (PedsQL) (Varni, Seid & Rode, 1999) will be used to measure child's health related quality of life during the past month. The scale measures child´s quality of health on four subscales namely, physical functioning, emotional functioning, social functioning and school functioning. The items are rated on 4 points Likert scale ranging from (1) 'no problem' to (4) 'almost always a problem'. Items are then reverse-scored and linearly transformed to a 0-100, so that higher scores indicate better quality of life. This tool yields a total score (all 23 items), physical health summary score (8 items), psycho-social health summary score (10 items) and school functioning score (5 items).
Pediatric Quality of Life (Peds-QL)-Family impact module | At baseline, immediate and 3-months' post-intervention.
  Peds-QL family impact module will be used to assess parents' health related quality of life. PedsQL family impact module is a 36-item scale that measures quality of life on 6 sub-scales namely; physical functioning, emotional functioning, social functioning, cognitive functioning, communication, worry, daily activities and family relationships. Items are rated on a 5-point Likert scale (0 = never to 4 = almost always). Total score is calculated by summing all 36 items divided by the number of items answered. The parent health related quality of life summary score (20 items) is computed as the sum of the items divided by the number of items answered in the physical, emotional, social, and cognitive functioning scales.
Alabama parenting scale | At baseline, immediate and 3- months' post-intervention.
  Alabama parenting scale will be used to measure parenting practices. Alabama parenting scale is a 42 item measure that encompasses five dimensions of parenting: (1) positive involvement with children, (2) supervision and monitoring, (3) use of positive discipline techniques, (4) consistency in the use of such discipline and (5) use of corporal punishment. Items are rated on a 5-point Likert scale (1 = never to 5 = almost always). Total score is calculated by summing all items.
Health Services Utilization: | At baseline and 3-months' post-intervention.
  The cost of health services utilization from the time proceeding assessment will be assessed with the adapted Client Services Receipt Inventory (CSRI). It has been adapted to use for the families of children with psycho-social distress. It measures the utilization of various health and social care services including time and opportunity losses by the families in the care of their child with psycho-social distress.
Short Warwick Edinburgh Wellbeing Scale (SWEWS) | At baseline, immediate and 3-months' post-intervention.
  The short version of the Warwick-Edinburgh Mental Well-being Scale will be used to evaluate the mental well-being of children. Statements of the measure are positively worded with five response categories from 'none of the time' to 'all of the time'. Children and young people are asked to describe their experiences over the past two weeks. Higher scores indicate higher positive mental well-being

CONTACTS AND LOCATIONS:
Overall Officials: Atif Rahman, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jellinek MS, Murphy JM, Burns BJ. Brief psychosocial screening in outpatient pediatric practice. J Pediatr. 1986 Aug;109(2):371-8. doi: 10.1016/s0022-3476(86)80408-5. PMID 3734977
- [Result] Dawson KS, Watts S, Carswell K, Shehadeh MH, Jordans MJD, Bryant RA, Miller KE, Malik A, Brown FL, Servili C, van Ommeren M. Improving access to evidence-based interventions for young adolescents: Early Adolescent Skills for Emotions (EASE). World Psychiatry. 2019 Feb;18(1):105-107. doi: 10.1002/wps.20594. No abstract available. PMID 30600639
- [Result] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Result] Thabane L, Hopewell S, Lancaster GA, Bond CM, Coleman CL, Campbell MJ, Eldridge SM. Methods and processes for development of a CONSORT extension for reporting pilot randomized controlled trials. Pilot Feasibility Stud. 2016 May 20;2:25. doi: 10.1186/s40814-016-0065-z. eCollection 2016. PMID 27965844
- [Derived] Hamdani SU, Huma ZE, Tamizuddin-Nizami A, Baneen UU, Suleman N, Javed H, Malik A, Wang D, Mazhar S, Khan SA, Minhas FA, Rahman A. Feasibility and acceptability of a multicomponent, group psychological intervention for adolescents with psychosocial distress in public schools of Pakistan: a feasibility cluster randomized controlled trial (cRCT). Child Adolesc Psychiatry Ment Health. 2022 Jun 21;16(1):47. doi: 10.1186/s13034-022-00480-z. PMID 35729589